CLINICAL TRIAL: NCT02974374
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Study To Assess Safety, Tolerability And Pharmacokinetics Of Single, Escalating, Oral Doses Of Pf-06835919 In Healthy Adult Subjects
Brief Title: Single Dose of PF-06835919 Escalation Study in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: C1061001
Record Dates: First submitted 2016-10-11; First posted 2016-11-28 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — PF-06835919

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- PF-06835919 (Experimental)
  Interventions: Drug: PF-06835919
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-06835919 — Single or repeated, escalating dose
  Arms: PF-06835919
Other: Placebo — Single or repeated, escalating dose
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and pharmacokinetics of a single dose of PF-06835919 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and female of non-childbearing potential;
* Body Mass Index 21.5 to 30.5 kg/m2 (inclusive);
* Total body weight >50 kg (110 lbs).

Exclusion Criteria:

-Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of Subjects experiencing an Adverse Event | Screening up to 28 days after last dose of study medication
  Assessment by adverse event monitoring, 12 lead ECGs, telemetry, vital signs and clinical safety laboratory measurements. Treatment-related AE was any untoward medical occurrence attributed to study drug in a subject who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Drug was assessed by the investigator (Yes/No). Subjects with multiple occurrences of an AE within a category were counted once within the category.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) for PF-06835919 | 0, 0.33, 1, 2, 3, 4, 5, 6, 8,10, 12, 16, 24, and 48 hours post dose
Time to Reach Maximum Observed Concentration for PF-06835919 | 0, 0.33, 1, 2, 3, 4, 5, 6, 8,10, 12, 16, 24, and 48 hours post dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-06835919 | 0, 0.33, 1, 2, 3, 4, 5, 6, 8,10, 12, 16, 24, and 48 hours post dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0- infinity)] for PF-06835919 | 0, 0.33, 1, 2, 3, 4, 5, 6, 8,10, 12, 16, 24, and 48 hours post dose
  AUC (0-infinity)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-infinity). It is obtained from AUC (0-t) plus AUC (t-infinity).
Plasma Decay Half-Life (t1/2) for PF-06835919 (as permitted) | 0, 0.33, 1, 2, 3, 4, 5, 6, 8,10, 12, 16, 24, and 48 hours post dose
  Plasma Decay Half-Life (t1/2)
Apparent Total Body Clearance (CL/F) for PF-06835919 (as permitted) | 0, 0.33, 1, 2, 3, 4, 5, 6, 8,10, 12, 16, 24, and 48 hours post dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after apparent total body clearance is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Apparent Volume of Distribution (Vz/F) for PF-06835919 (as permitted) | 0, 0.33, 1, 2, 3, 4, 5, 6, 8,10, 12, 16, 24, and 48 hours post dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C1061001&StudyName=A+Phase+1%2C+Randomized%2C+Double-blind%2C+Placebo+Controlled+Study+To+Assess+Safety%2C+Tolerability+And+Pharmacokinetics+Of+Single%2C+Escalating%2C+Oral+Doses+Of+Pf-06835919+In+Healthy+Adult+Subjects
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C1061001&StudyName=A+Phase+1%2C+Randomized%2C+Double-blind%2C+Placebo-controlled+Study+To+Assess+Safety%2C+Tolerability+And+Pharmacokinetics+Of+Single%2C+Escalating%2C+Oral+Doses+Of+Pf-06835919+In+Healthy+Adult+Subjects